CLINICAL TRIAL: NCT03306784
Title: Transversal Study of Correlations Between Pain Catastrophizing Scale (PCS) and RAPID3 Score According to Ten Categories of Conditions Seen in an Outpatient Rheumatology Clinic
Brief Title: Pain Catastrophizing and Routine Assessment of Patient Index Data 3(RAPID3) in Ten Categories of Rheumatology Outpatients
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0182
Record Dates: First submitted 2017-07-05; First posted 2017-10-11 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Arthritis, Rheumatoid; Spondyloarthritis; Inflammatory Rheumatisms; Systemic Disorders
Keywords: RAPID3; pain catastrophizing
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Rheumatic Fever | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaires — questionnaires, including RAPID3 and pain catastrophizing scales

SUMMARY:
Fulfilling by all patients consequently seen by 6 rheumatologists in a same outpatient rheumatology clinic (in at least one month period) of a set of 6 questionnaires, including RAPID3 and pain catastrophizing scales.

DETAILED DESCRIPTION:
Fulfilling by all patients (seen by 6 rheumatologists in a same outpatient rheumatology clinic from a university French hospital in at least one month period) of a set of 6 questionnaires including a RAPID3 score (Routine Assessment of Patient Index Data 3) and pain catastrophizing scale, as well as Pain detect and Hospital Anxiety and Depression scale questionnaires (HAD) , in ten predefined categories of disorders: rheumatoid arthritis; any spondyloarthritis; other inflammatory rheumatisms or systemic disorders; osteoarthritis of the upper part of the body; osteoarthritis of the lower part of the body; back pain and/or radiculalgia; bone disorders, including osteoporosis; tendinosis and other soft tissue conditions; peripheral neuropathy, including entrapment neuropathies; fibromyalgia and related conditions.

ELIGIBILITY:
Inclusion Criteria:

* any outpatient aged 18 or more, agreeing to fulfil the set of 6 questionnaires
* Man or woman coming to the Rheumatology Department of the Nantes University Hospital with a senior rheumatologist

Exclusion Criteria:

* Patients not fluent enough in French or suffering from neurological or psychological disorders making their responses unreliable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 Men or women coming to the Rheumatology Department of the Nantes University Hospital with a senior rheumatologist agreeing to fulfil the set of 6 questionnaires
Sampling Method: Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Ranking of PCS scores according to the underlying disorders (10 predefined categories), and also ranking of RAPID-3 scores according to the underlying disorders (10 predefined categories). | At least one month for each physician, and at least 30 patients in each category (whatever the physician seen).
  Composite score: RAPID3 (0-30) and PCS (0-52) are widely used scales, suitable for routine fulfillment by outpatients.

SECONDARY OUTCOMES:
Ranking of correlations between RAPID3 and Pain catastrophizing scale (PCS) (13 items) scores in the 10 subsets of categories listed above (from the strongest correlation to the lowest correlation) | At least one month for each physician, and at least 30 patients in each category (whatever the physician seen).
  RAPID3 (0-30) and PCS (0-52) are widely used scales, suitable for routine fulfillment by outpatients

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Berthelot, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France